CLINICAL TRIAL: NCT03765632
Title: Efficacy and Safety of a Cryopreserved Formulation of Autologous CD34+ Haematopoietic Stem Cells Transduced ex Vivo With Elongation Factor 1α Short Form (EFS) Lentiviral Vector Encoding for Human ADA Gene in Subjects With Severe Combined Immunodeficiency (SCID) Due to Adenosine Deaminase Deficiency
Brief Title: Efficacy and Safety of the Cryopreserved Formulation of OTL-101 in Subjects With ADA-SCID
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: Orchard Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTL-101-5; 17IC04 (Other: UCL Great Ormond Street Institute of Child Health)
Record Dates: First submitted 2018-08-08; First posted 2018-12-05 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Severe Combined Immunodeficiency Due to ADA Deficiency
Keywords: Gene therapy; Hematopoietic stem and progenitor cells; Lentiviral vector; ADA-SCID
MeSH Terms: conditions — Severe combined immunodeficiency due to adenosine deaminase deficiency | interventions — Busulfan; pegademase bovine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gene Therapy (Experimental): Infusion of autologous cryopreserved EFS-ADA LV CD34+ cells
  Interventions: Genetic: Infusion of autologous cryopreserved EFS-ADA LV CD34+ cells (OTL-101); Drug: Busulfan; Drug: Peg-Ada

INTERVENTIONS:
Genetic: Infusion of autologous cryopreserved EFS-ADA LV CD34+ cells (OTL-101) — Autologous cryopreserved EFS-ADA LV CD34+ cells (OTL-101) are infused intravenously
  Other Names: OTL-101
Drug: Busulfan — Busulfan is used for non-myeloablative conditioning
Drug: Peg-Ada — Peg-Ada Enzyme Replacement Therapy (ERT) is discontinued at Day +30 (-3/+15 days) after successful engraftment

SUMMARY:
This is a prospective, non-randomized, single-cohort, longitudinal, single-center, clinical study designed to assess the efficacy and safety of a cryopreserved formulation of OTL-101 (autologous CD34+ hematopoietic stem/progenitor cells transduced ex vivo with EFS (Elongation Factor 1α Short form) Lentiviral Vector (LV) encoding for the human ADA gene) administered to ADA-SCID subjects between the ages of >/=30 days and <18 years of age, who are not eligible for an Human Leukocyte Antigen (HLA) matched sibling/family donor and meeting the inclusion/exclusion criteria. The OTL-101 product is infused after a minimal interval of at least 24 hours following the completion of reduced intensity conditioning. For subjects who successfully receive the OTL-101 product, pegademase bovine (PEG-ADA) Enzyme Replacement Therapy (ERT) is discontinued at Day+30 (-3/+15) after the transplant. After their discharge from hospital, the subjects will be seen at regular intervals to review their history, perform examinations and draw blood samples to assess immunity and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent prior to any study related procedures. In this study consent must be provided by the parents/legal guardians and, where applicable according to local laws, a signed assent from the child
2. Subjects ≥30 days and <18 years of age,
3. With a diagnosis of ADA-SCID based on:

   1. . Evidence of ADA deficiency, defined as: i. Decreased ADA enzymatic activity in erythrocytes, leukocytes, skin fibroblasts, or in cultured foetal cells to levels consistent with ADA-SCID as determined by the reference laboratory, or ii. Identified mutations in ADA alleles consistent with a severe reduction in ADA activity,
   2. . Evidence of ADA-SCID based on either: i. Family history of a first order relative with ADA deficiency and clinical and laboratory evidence of severe immunologic deficiency, or ii. Evidence of severe immunologic deficiency in subjects prior to the institution of immune restorative therapy, based on

   Lymphopenia (absolute lymphocyte count <400 cells/mL) OR absence or low number of T-cells (absolute CD3+ count < 300 cells/mL), or

   Severely decreased T lymphocyte blastogenic responses to phytohemagglutinin (either <10% of lower limit of normal controls for the diagnostic laboratory, or <10% of the response of the normal control of the day, or stimulation index <10), or

   Identification of SCID by neonatal screening revealing low T cell Receptor Excision Circle (TREC) levels.
4. Ineligible for or with no available matched family donor for allogeneic Bone Marrow (BM) transplantation, defined as the absence of a medically eligible HLA-identical sibling or family donor, with normal immune function, who could serve as an allogeneic bone marrow donor.
5. Females of child-bearing age will be required to provide a negative pregnancy test 30 days prior to Visit 2.
6. Subjects and their parents/legal guardians must be willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study period and willing to return to the clinic for the follow up evaluation as specified in the protocol.

Exclusion Criteria:

1. Ineligible for autologous hematopoietic stem cell (HSC) procedure.
2. Other conditions which in the opinion of the Principal Investigator and/or Co-Investigators, contraindicate the harvest of bone marrow, the administration of Busulfan and the infusion of transduced cells, or which indicate an inability of the subject or subject's parent/legal guardian to comply with the protocol.
3. Haematologic abnormality, defined as:

   Anaemia (Hb <8.0 g/dl). Evidence of bi/trilineage cytopaenia (haemoglobin <8 g/dl, neutrophils <0.5 x 109/L, platelets 50 x 109/L). Thrombocytopaenia (platelet count <50,000/mm3). Prothrombin time or partial thromboplastin time (PTT) >2 x upper limit of normal (ULN) (subjects with a correctable deficiency controlled on medication will not be excluded).
   * Cytogenetic abnormalities of Peripheral Blood (PB), BM or amniotic fluid (if available). If cytogenetic testing has not been performed on cells from amniocentesis, assessment should be by karyotype, Comparative genomic hybridization (CGH), and or whole exome sequencing (WES).
   * Prior allogeneic HSC transplant (HSCT) with cytoreductive conditioning.
4. Pulmonary abnormality, defined as:

   * Resting O2 saturation by pulse oximetry <90% on room air.
   * Chest X-ray indicating active or progressive pulmonary disease. Note: Chest X-ray indicating residual signs of treated pneumonitis is acceptable for eligibility.
5. Cardiac abnormality, defined as:

   * Abnormal ECG indicating cardiac pathology.
   * Uncorrected congenital cardiac malformation with clinical symptoms.
   * Active cardiac disease, including clinical evidence of congestive heart failure, cyanosis, hypotension.
   * Poor cardiac function as evidenced by left ventricular ejection fraction <40% on echocardiogram.
6. Neurologic abnormality, defined as:

   * Significant neurologic abnormality revealed by examination.
   * Uncontrolled seizure disorder.
7. Known history of significant renal abnormality.
8. Known history of significant hepatic or gastrointestinal abnormality.
9. Oncologic disease, defined as:

   * Evidence of active malignant disease other than Dermatofibrosarcoma Protuberans( DFSP) 2.
   * Evidence of DFSP expected to require anti-neoplastic therapy within the 5 years following the infusion of genetically corrected cells (if anti-neoplastic therapy has been completed, a subject with a history of DFSP can be included).
   * Evidence of DFSP expected to be life-limiting within the 5 years following the infusion of genetically corrected cells.
10. Known sensitivity to Busulfan.
11. Confirmation of an infectious disease by deoxyribonucleic acid (DNA) polymerase chain reactions (PCR) positive at time of screening assessment according to local protocols/procedures (including HIV-1 and hepatitis B).
12. The subject is pregnant or has a major congenital anomaly.
13. Is likely to require treatment during the study with drugs that are not permitted by the study protocol.
14. The subject has previously received another form of gene therapy.

Ages: 30 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Overall survival at 12 months post OTL-101 infusion | 12 Months
  Overall survival is defined as the proportion of subjects alive
Event free survival at 12 months post OTL-101 infusion | 12 Months
  Event-free survival is defined as the proportion of subjects alive with no "event", an "event" being the resumption of Peg-Ada ERT or the need for a rescue stem cell transplant (SCT), or death

SECONDARY OUTCOMES:
Overall survival at 24 months post OTL-101 infusion | 24 months
  Overall survival is defined as the proportion of subjects alive
Event free survival at 24 months post OTL-101 infusion | 24 Months
  Event-free survival is defined as the proportion of subjects alive with no "event", an "event" being the resumption of Peg-Ada ERT or the need for a rescue stem cell transplant (SCT), or death
Safety evaluation including infection rates | 12 and 24 months
Safety evaluation including performance outcomes | 12 and 24 months
Safety evaluation including immune reconstitution | 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Claire Booth, Dr, Principal Investigator — Great Ormond Street Hospital NHS Foundation Trust
Locations (1):
- Great Ormond Street Hospital for Children NHS Foundation Trust, London, United Kingdom